CLINICAL TRIAL: NCT06698016
Title: A Study to Evaluate the Effect of Multiple Oral Doses of Efavirenz on the Single-Dose Pharmacokinetics of Nemtabrutinib in Healthy Participants
Brief Title: A Study of the Effect of Efavirenz on the Plasma Levels of Nemtabrutinib (MK-1026-014)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 1026-014
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — ARQ531; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Period 1: Nemtabrutinib (Experimental): Participants receive a single dose of nemtabrutinib followed by a protocol specified wash-out period.
  Interventions: Drug: Nemtabrutinib
- Period 2: Nemtabrutinib + Efavirenz (Experimental): Participants receive oral doses of efavirenz once daily on Days 1 to 24 with a single oral dose of nemtabrutinib given with efavirenz on Day 11.
  Interventions: Drug: Nemtabrutinib; Drug: Efavirenz

INTERVENTIONS:
Drug: Nemtabrutinib — Oral administration
  Other Names: MK-1026; ARQ 531
Drug: Efavirenz — Oral administration
  Arms: Period 2: Nemtabrutinib + Efavirenz

SUMMARY:
The goal of the study is to learn what happens to levels of nemtabrutinib (MK-1026) in a healthy person's body over time. Researchers will compare what happens to nemtabrutinib in the body when it is given with or without another medicine called efavirenz.

ELIGIBILITY:
Inclusion Criteria

The key inclusion criteria include but are not limited to the following:

* Is in good health based on medical history, physical examination, vital sign (VS) measurements, electrocardiograms (ECGs) and laboratory safety tests performed before allocation
* Has a body mass index (BMI) > 18 kg/m2 and ≤ 32 kg/m^2

Exclusion Criteria

The key exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has a history of cancer (malignancy)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Nemtabrutinib | Predose and at designated time points (up to 2 weeks)
  Blood samples will be collected to determine the AUC0-inf of nemtabrutinib.

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to 24 hours (AUC0-24hrs) of Nemtabrutinib | Predose and at designated time points (up to 24 hours postdose)
  Blood samples will be collected to determine the AUC0-24hr of nemtabrutinib.
Maximum Plasma Concentration (Cmax) of Nemtabrutinib | Predose and at designated time points (up to 2 weeks)
  Blood samples will be collected to determine the Cmax of nemtabrutinib.
Time to Maximum Plasma Concentration (Tmax) of Nemtabrutinib | Predose and at designated time points (up to 2 weeks postdose)
  Blood samples will be collected to determine the Tmax of nemtabrutinib.
Apparent Clearance (CL/F) of Nembrutinib | Predose and at designated time points (up to 2 weeks)
  Blood samples will be collected to determine the CL/F of nemtabrutinib.
Apparent Volume of Distribution During Terminal Phase (Vz/F) Nemtabrutinib | Predose and at designated time points (up to 2 weeks)
  Blood samples will be collected to determine the Vz/F of nemtabrutinib.
Apparent Terminal Half-life (t1/2) of Nemtabrutinib | Predose and at designated time points (up to 2 weeks)
  Blood samples will be collected to determine the t1/2 of nemtabrutinib.
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 2 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 2 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharpe & Dohme LLC
Locations (1):
- Altasciences Clinical Kansas, Inc. (Site 0001), Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/